CLINICAL TRIAL: NCT01010282
Title: Safety and Efficacy of Two Artificial Tears in Dry Eye Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: AG9965-002
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Results first posted 2011-12-13 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-07

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Glycerol; Polysorbates

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Glycerin and Polysorbate 80 based artificial tear (Active Comparator): Glycerin and Polysorbate 80 based artificial tear
  Interventions: Drug: Glycerin and Polysorbate 80 based artificial tear
- Artificial Tears Formulation 1 (Experimental): Formulation 1: Carboxymethylcellulose sodium, glycerin and Polysorbate 80, based artificial tear
  Interventions: Drug: Formulation 1: Carboxymethylcellulose sodium, glycerin and Polysorbate 80, based artificial tear
- Artificial Tears Formulation 2 (Experimental): Formulation 2: Carboxymethylcellulose sodium, glycerin, and Polysorbate 80 based artificial tear
  Interventions: Drug: Formulation 2: Carboxymethylcellulose sodium, glycerin, and Polysorbate 80 based artificial tear

INTERVENTIONS:
Drug: Glycerin and Polysorbate 80 based artificial tear — 1-2 drops in each eye, as needed, but at least twice daily
  Other Names: Refresh Dry Eye Therapy® Lubricant Eye Drops
  Arms: Glycerin and Polysorbate 80 based artificial tear
Drug: Formulation 1: Carboxymethylcellulose sodium, glycerin and Polysorbate 80, based artificial tear — 1-2 drops in each eye, as needed, but at least twice daily
  Arms: Artificial Tears Formulation 1
Drug: Formulation 2: Carboxymethylcellulose sodium, glycerin, and Polysorbate 80 based artificial tear — 1-2 drops in each eye, as needed, but at least twice daily
  Arms: Artificial Tears Formulation 2

SUMMARY:
This study will evaluate the safety, efficacy, and acceptability of two artificial tears compared to a currently available artificial tear in subjects with dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Current use of an artificial tear at least twice daily, for at least three months prior to Day 1, on average
* Ability/agreement to wear habitual correction (glasses) during study period

Exclusion Criteria:

* Known allergy or sensitivity to the study product(s) or its components
* Anticipate contact lens wear during the study, or subject has worn contact lenses in the last six months
* Chronic use of systemic medications which may affect a dry eye condition
* Active ocular allergy or infection
* Use of Restasis® or other topical cyclosporine products within 3 months prior to Day 1
* Current use of any topical ophthalmic medications, have used within 2 weeks prior to Day 1, or are likely to use during study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- San Diego, California, United States

REFERENCES:
- [Derived] Simmons PA, Carlisle-Wilcox C, Chen R, Liu H, Vehige JG. Efficacy, safety, and acceptability of a lipid-based artificial tear formulation: a randomized, controlled, multicenter clinical trial. Clin Ther. 2015 Apr 1;37(4):858-68. doi: 10.1016/j.clinthera.2015.01.001. Epub 2015 Feb 4. PMID 25659956

RESULTS

PARTICIPANT FLOW:
Groups:
- Artificial Tears Formulation 1: Artificial Tears Formulation 1
- Artificial Tears Formulation 2: Artificial Tears Formulation 2
Period: Overall Study
Arm/Group | Artificial Tears Formulation 1 | Artificial Tears Formulation 2 | Glycerin and Polysorbate 80 Based Artificial Tear
Started | 97 | 95 | 96
Completed | 91 | 88 | 77
Not Completed | 6 | 7 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Artificial Tears Formulation 1 | Artificial Tears Formulation 2 | Glycerin and Polysorbate 80 Based Artificial Tear | Total
Number analyzed (Participants) | 97 | 95 | 96 | 288
Age, Customized [Number; unit: participants]
  <30 years | 6 | 9 | 4 | 19
  between 30 and 40 years | 6 | 9 | 11 | 26
  >40 years | 85 | 77 | 81 | 243
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 70 | 70 | 216
  Male | 21 | 25 | 26 | 72

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Subjective Evaluation of Symptom of Dryness (SESoD)Score at Day 90
Description: Change from baseline in SESoD score at day 90. The SESoD is a 5-point scale where 0 equals no dryness, 1 equals trace dryness, 2 equals mild dryness, 3 equals moderate dryness, and 4 equals severe dryness. A negative number change from baseline indicates a decrease (improvement) in the symptom of dryness.
Time Frame: Baseline (Day 1), Day 90
Population: Intent-to-treat, which includes all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Artificial Tears Formulation 1 | Artificial Tears Formulation 2 | Glycerin and Polysorbate 80 Based Artificial Tear
Number analyzed (Participants) | 97 | 95 | 96
Scores on a Scale
  Baseline (Day 1) | 2.7 (0.59) | 2.8 (0.67) | 2.8 (0.65)
  Change from Baseline at Day 90 | -0.7 (0.89) | -0.7 (0.90) | -0.7 (0.96)

2. Secondary Outcome: Change From Baseline in the Ocular Surface Disease Index (OSDI) Total Score at Day 90
Description: Change from baseline in the OSDI total score at day 90. The OSDI is a 12-question survey for patients to document their dry eye disease symptoms. The OSDI consists of a 5-point scale (0=none of the time and 4=all of the time), with higher scores representing greater disability. The scores are totaled over the 12 questions and converted to a score of 0-100 (0=no disability and 100=complete disability). A negative number change from baseline represents an improvement.
Time Frame: Baseline (Day 1), Day 90
Population: Intent-to-treat, which includes all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Artificial Tears Formulation 1 | Artificial Tears Formulation 2 | Glycerin and Polysorbate 80 Based Artificial Tear
Number analyzed (Participants) | 97 | 95 | 96
Scores on a Scale
  Baseline (Day 1) | 33.6 (20.19) | 35.1 (19.18) | 37.3 (18.67)
  Change from Baseline at Day 90 | -7.2 (19.47) | -10.6 (18.43) | -9.1 (19.68)

3. Secondary Outcome: Change From Baseline in Tear Break-up Time (TBUT) at Day 90
Description: Change from baseline in TBUT at day 90. TBUT is the time required for dry spots to appear on the surface of the eye after blinking. The longer it takes, the more stable the tear film. A short TBUT is a sign of poor tear film. A positive number change from baseline indicates an increase in TBUT (improvement).
Time Frame: Baseline (Day 1), Day 90
Population: Intent-to-treat, which includes all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Artificial Tears Formulation 1 | Artificial Tears Formulation 2 | Glycerin and Polysorbate 80 Based Artificial Tear
Number analyzed (Participants) | 97 | 95 | 96
Seconds
  Baseline (Day 1) | 4.90 (1.768) | 5.04 (1.653) | 5.09 (1.782)
  Change from Baseline at Day 90 | 1.49 (2.955) | 2.02 (3.812) | 1.81 (3.464)

4. Secondary Outcome: Change From Baseline in Corneal Staining at Day 90
Description: Change from baseline in corneal staining at day 90. The cornea is the transparent front part of the eye which covers the iris and pupil. Corneal staining following administration of fluorescein dye in the eye is graded using a 6-point scale (0=no staining, 5=severe staining) over 5 areas of the clear central part of the eye for a minimum score of 0 and maximum score of 25. The higher the grade score, the worse the dry eye condition. A negative number change from baseline represents a decrease in corneal staining (improvement).
Time Frame: Baseline (Day 1), Day 90
Population: Intent-to-treat, which includes all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Artificial Tears Formulation 1 | Artificial Tears Formulation 2 | Glycerin and Polysorbate 80 Based Artificial Tear
Number analyzed (Participants) | 97 | 95 | 96
Scores on a scale
  Baseline (Day 1) | 4.2 (3.14) | 4.2 (2.91) | 4.5 (3.15)
  Change from Baseline at Day 90 | 0.2 (3.35) | -0.5 (3.01) | 0.8 (4.14)

5. Secondary Outcome: Change From Baseline in Conjunctival Staining Severity Score at Day 90
Description: Change from baseline in conjunctival staining severity score at day 90. The conjunctiva is the clear membrane covering the white surface of the eye. Conjunctival staining following ocular administration of lissamine green dye was graded using a 6-point scale (0=no staining, 5=severe staining) over 6 areas of the white part of the eye for a minimum score of 0 and a maximum score of 30. The higher the score, the worse the dry eye condition. A negative number change from baseline represents a decrease in the severity of conjunctival staining (improvement).
Time Frame: Baseline (Day 1), Day 90
Population: Intent-to-treat, which includes all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Artificial Tears Formulation 1 | Artificial Tears Formulation 2 | Glycerin and Polysorbate 80 Based Artificial Tear
Number analyzed (Participants) | 97 | 95 | 96
Scores on a scale
  Baseline (Day 1) | 5.1 (4.71) | 4.9 (4.37) | 5.2 (4.95)
  Change from Baseline at Day 90 | -0.5 (4.17) | -0.7 (4.53) | -0.7 (3.89)

ADVERSE EVENTS:
Arm/Group | Artificial Tears Formulation 1 | Artificial Tears Formulation 2 | Glycerin and Polysorbate 80 Based Artificial Tear
Serious Adverse Events (participants affected / at risk) | 2/97 | 0/95 | 4/96
Other Adverse Events (participants affected / at risk) | 28/97 | 14/95 | 37/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Artificial Tears Formulation 1 (N=97) | Artificial Tears Formulation 2 (N=95) | Glycerin and Polysorbate 80 Based Artificial Tear (N=96)
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Artificial Tears Formulation 1 (N=97) | Artificial Tears Formulation 2 (N=95) | Glycerin and Polysorbate 80 Based Artificial Tear (N=96)
Visual acuity reduced (Eye disorders) | 16 | 7 | 11
Vision blurred (Eye disorders) | 5 | 3 | 7
Eye pain (Eye disorders) | 3 | 1 | 6
Photophobia (Eye disorders) | 3 | 1 | 5
Instillation site pain (General disorders) | 1 | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo